CLINICAL TRIAL: NCT04616469
Title: Evaluation of the Effect of Root Canal Shaping With TruNatomy on Postoperative Pain and Operative Torque Generated During Instrumentation: A Randomized Clinical Trial
Brief Title: Evaluation of the Effect of Root Canal Shaping With TruNatomy on Postoperative Pain and Operative Torque Generated During Instrumentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tarek Ali El Mosalamy, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO:3-3-5 (8-10-2020)
Record Dates: First submitted 2020-10-08; First posted 2020-11-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal treatment using RaCe rotary system (Active Comparator): Canal shaping using RaCe rotary system powered with endodontic motor with real time torque monitoring capacity
  Interventions: Procedure: Root canal treatment using race rotary instruments
- Root canal treatment using TruNatomy rotary system (Experimental): Canal shaping using TruNatomy rotary system powered with endodontic motor with real time torque monitoring capacity
  Interventions: Procedure: Root canal treatment using TruNaomy rotary files

INTERVENTIONS:
Procedure: Root canal treatment using TruNaomy rotary files — Trunatomy rotary files will be used for the process of cleaning and shaping of the root canal system
  Arms: Root canal treatment using TruNatomy rotary system
Procedure: Root canal treatment using race rotary instruments — Race rotary files will be used for the process of cleaning and shaping of the root canal system
  Arms: Root canal treatment using RaCe rotary system

SUMMARY:
The aim of the present study is to compare the effect of canal shaping using TruNatomy and RaCe rotary systems in bi-rooted maxillary premolars in terms of:

* Post operative pain: incidence and intensity
* Real time torque generated during mechanical instrumentation using real time torque motoring endodontic motor
* Time needed for the instruments to reach to the full working length

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition and no contributory systemic disease.
* Age between 30-60 years old.
* Males & Females.
* Patients' acceptance for participating in the trial through an informed consent
* Maxillary permanent premolar teeth:

  * Diagnosed clinically and radiographically with pulp necrosis
  * With or without periapical radiolucency
  * Negative response of pulp tissue to thermal and electric pulp tester
  * Possessing two independent roots each having a type I canal
  * Patent canals with no internal calcification or resorptive lesions
  * Fully formed roots
  * Root curvatures less than 30

Exclusion Criteria:

* Patient with contributory medical condition
* Badly destructed teeth
* Patients with pre-operative pain
* Patients having significant systemic disorders
* Patients with two or more adjacent teeth requiring root canal therapy
* Patients who had received antibiotics in the last month
* Teeth presenting with:

  * Positive response to thermal or electric pulp tester
  * History of trauma or previous endodontic treatment
  * Immature or open apices
  * Association with acute periapical abscess and swelling or fistulous tract
  * Fused roots at any level
  * Canals larger than size 15# K-file
  * Periodontonal/ endodontic lesions
  * Mobility higher than grade I
  * Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.
  * Severe root curvature (>30)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain using visual analogue scale | at 24 hours post treatment
  pain after treatment would be measured with a VAS scale from 0-10 cm with zero representing the least amount of pain and 10 representing the worst pain possible
Post operative pain using visual analogue scale | at 48 hours post treatment
  pain after treatment would be measured with a VAS scale from 0-10 cm with zero representing the least amount of pain and 10 representing the worst pain possible
Post operative pain using visual analogue scale | at 72 hours post treatment
  pain after treatment would be measured with a VAS scale from 0-10 cm with zero representing the least amount of pain and 10 representing the worst pain possible
Post operative pain using visual analogue scale | at 1 week post treatment
  pain after treatment would be measured with a VAS scale from 0-10 cm with zero representing the least amount of pain and 10 representing the worst pain possible

SECONDARY OUTCOMES:
operative torque generated during instrumentation | during treatment
  real time operative torque exerted on the instrument through out the shaping process and until the instrument reaches the full working length will be measured using a torque measuring motor in real time
time required for the instrument to reach the full working length | during treatment
  time required for the the instrument to reach the full length and complete the shaping process will be calculated using a Realtime torque motoring motor

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gambarini G, Galli M, Seracchiani M, Di Nardo D, Versiani MA, Piasecki L, Testarelli L. In Vivo Evaluation of Operative Torque Generated by Two Nickel-Titanium Rotary Instruments during Root Canal Preparation. Eur J Dent. 2019 Oct;13(4):556-562. doi: 10.1055/s-0039-1698369. Epub 2019 Dec 31. PMID 31891973
- [Background] Zand V, Milani AS, Hassani Dehkharghani A, Rahbar M, Tehranchi P. Treatment of Necrotic Teeth Using Two Engine-Driven Systems and Patient's Postoperative Pain: A Double-Blind Clinical Trial. Iran Endod J. 2016 Fall;11(4):267-272. doi: 10.22037/iej.2016.3. PMID 27790254
- [Derived] Al-Mosalmy TA, El-Far HM, Gomaa MM, Morsy DA. Impact of root canal shaping using TruNatomy on postoperative pain and operative torque generation: a randomized clinical trial. BMC Oral Health. 2025 Jul 19;25(1):1222. doi: 10.1186/s12903-025-06418-z. PMID 40684114